CLINICAL TRIAL: NCT03504007
Title: Standardized, Guidelines Directed But Patients Oriented Clinical Practice Prospectively Registered
Brief Title: Registry of Patients Prescribed Anticoagulation
Acronym: STAGPOR
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Damon E. Houghton, Principal Investigator, Mayo Clinic
Other Study IDs: 13-001404
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Acute Deep Vein Thrombosis; Acute Pulmonary Embolism
Keywords: Deep Vein Thrombosis; Pulmonary Embolism; Apixaban; Rivaroxaban; Dabigatran; Edoxaban
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Gonda Vascular Center- Thrombophilia Clinic at Mayo Clinic in Rochester, Minnesota utilizes a standardized, guideline-directed, yet patient-oriented approach for treating patients diagnosed with venous thromboembolism (VTE).This study is the ongoing registry of clinical practice with standardized approach to patient assessment and therapy. As most of registries it does not have any definite number of recruited subjects or the date of study completion but provides anticipated number of recruited subjects and the time of anticipated enrolment which was provided only because of formal requirement related to structure of ClinicalTrials.gov website. This number will be updated and upgraded as we continue this registry.

The rates of VTE recurrence, major bleeding, clinically relevant non-major bleeding (CRNMB) and survival in patients treated with anticoagulation for acute VTE are assessed during prospective observation. VTE cases include an acute deep vein thrombosis (DVT) of lower or upper extremities, splanchnic veins, gonadal, renal, cerebral veins thrombosis and pulmonary embolism (PE). Therapy includes the whole spectrum of FDA approved anticoagulants such as "classic" agents: warfarin and heparinoids and the newer direct oral anticoagulants (DOACs) such as rivaroxaban, dabigatran, apixaban, and edoxaban.

DETAILED DESCRIPTION:
When a patient has positive testing for acute VTE the radiologist interpreting the study contacts the Thrombophilia Center and the patient is immediately evaluated. Standardized information about guidelines endorsed anticoagulation therapy is provided in a uniform fashion with a standardized script for providers and a short summary table for the patient. This initial review also includes patient-specific cost information by contacting a pharmacy service phone-line. Patients with cancer-related VTE are counselled regarding the guideline endorsed use of low molecular heparin (LMWH) as the preferred option of anticoagulation and available data on DOACs. After the shared decision making is complete, the prescription is promptly filled at the pharmacy located within the same building, with the first dose administered within the ensuing hour. For patients with acute VTE diagnosed after hours, evaluation is accomplished in the Emergency Department; one dose of LMWH is administered and the patient is referred the next day to the Thrombophilia Clinic.

Patients with symptomatic PE or extensive symptomatic iliofemoral DVT are referred for prompt hospitalization. While in the hospital, they are consulted by a Vascular Medicine service and an appropriate follow up visit at the Thrombophilia Clinic is arranged. For patients with asymptomatic or minimally symptomatic pulmonary embolism (simplified Pulmonary Embolism Severity Index (PESI) score of 0), outpatient management is offered. All patients with cancer-associated PE are referred for lower extremity duplex ultrasound, and if symptomatic or if a central venous catheter is in place, also for upper extremity venous assessment.

Demographic and clinical data are entered into a REDCap. The registry is maintained on institutional servers, which are backed-up nightly and protected in controlled computer room with uninterrupted power supplies, data will never reside on a desktop computer system. Transfer of registry data will occur inside the Mayo Clinic firewall via our integrated high speed network. Analysis will be done using the most current version of SAS® software.

At the most recent update, over 2775 patients were enrolled. These data are used to analyze currently relevant clinical questions and are presented and published.

ELIGIBILITY:
Inclusion Criteria:

• VTE seen at Thrombophilia Clinic and treatment with anti-coagulant is started within 14 days of VTE diagnosis date.

Exclusion Criteria:

* Patients already on anticoagulation for other reasons or enrolled into anticoagulation clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic patients prescribed anticoagulation for treatment of acute DVT or PE. Treatment with all FDA-approved anticoagulants are captured in the database
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-03-01 (Actual); Primary Completion 2033-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of symptomatic, recurrent VTE. Incidence of major bleeding | 10 years
  Recurrent VTE clearly new compared to previous VTE. Major bleeding by ISTH definition

CONTACTS AND LOCATIONS:
Overall Officials: Damon Houghton, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janczak DT, Mimier MK, McBane RD, Kamath PS, Simmons BS, Bott-Kitslaar DM, Lenz CJ, Vargas ER, Hodge DO, Wysokinski WE. Rivaroxaban and Apixaban for Initial Treatment of Acute Venous Thromboembolism of Atypical Location. Mayo Clin Proc. 2018 Jan;93(1):40-47. doi: 10.1016/j.mayocp.2017.10.007. Epub 2017 Dec 6. PMID 29217335
- [Background] Bott-Kitslaar DM, Saadiq RA, McBane RD, Loprinzi CL, Ashrani AA, Ransone TR, Wolfgram AA, Berentsen MM, Wysokinski WE. Efficacy and Safety of Rivaroxaban in Patients with Venous Thromboembolism and Active Malignancy: A Single-Center Registry. Am J Med. 2016 Jun;129(6):615-9. doi: 10.1016/j.amjmed.2015.12.025. Epub 2016 Jan 18. PMID 26797081
- [Background] Houghton DE, Vlazny DT, Casanegra AI, Brunton N, Froehling DA, Meverden RA, Hodge DO, Peterson LG, McBane RD, Wysokinski WE. Bleeding in Patients With Gastrointestinal Cancer Compared With Nongastrointestinal Cancer Treated With Apixaban, Rivaroxaban, or Enoxaparin for Acute Venous Thromboembolism. Mayo Clin Proc. 2021 Nov;96(11):2793-2805. doi: 10.1016/j.mayocp.2021.04.026. Epub 2021 Aug 20. PMID 34425962
- [Background] Wysokinski WE, Froehling DA, Houghton DE, McBane RD, Vlazny DT, Bott-Kitslaar DM, Kuczmik W, Sutkowska K, Bator K, Hodge DO, Peterson LG, Casanegra AI. Effectiveness and safety of apixaban and rivaroxaban for acute venous thromboembolism therapy in patients with extremes in bodyweight. Eur J Haematol. 2020 Oct;105(4):484-494. doi: 10.1111/ejh.13471. Epub 2020 Jul 27. PMID 32557773
- [Background] Houghton DE, Casanegra AI, Peterson LG, Cochuyt J, Hodge DO, Vlazny D, McBane RD, Froehling D, Wysokinski WE. Treatment of upper extremity deep vein thrombosis with apixaban and rivaroxaban. Am J Hematol. 2020 Jul;95(7):817-823. doi: 10.1002/ajh.25820. Epub 2020 Apr 20. PMID 32267011
- [Derived] Hirao-Try Y, Vlazny DT, Meverden R, Houghton DE, Casanegra AI, Froehling DA, Hodge DO, Peterson LG, McBane RD, Wysokinski WE. Single versus multiple and incidental versus symptomatic subsegmental pulmonary embolism: clinical characteristics and outcome. J Thromb Thrombolysis. 2022 Jul;54(1):82-90. doi: 10.1007/s11239-021-02623-z. Epub 2022 Jan 7. PMID 34993715
- [Derived] Cambron JC, Saba ES, McBane RD, Casanegra AI, Villarraga HR, Houghton DE, Vlazny DT, Froehling D, Hodge D, Peterson LG, Bott-Kitslaar DM, Wysokinski WE. Adverse Events and Mortality in Anticoagulated Patients with Different Categories of Pulmonary Embolism. Mayo Clin Proc Innov Qual Outcomes. 2020 Jun 5;4(3):249-258. doi: 10.1016/j.mayocpiqo.2020.02.002. eCollection 2020 Jun. PMID 32542216
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials